CLINICAL TRIAL: NCT03377478
Title: Expanding the Pool in Lung Transplantation: The Use of Hepatitis C Positive Donor Lungs in Hepatitis C Negative Recipients
Brief Title: Expanding the Pool in Lung Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pablo Sanchez (Other)
Responsible Party: Sponsor-Investigator, Pablo Sanchez, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19030435
Record Dates: First submitted 2017-12-14; First posted 2017-12-19 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Hepatitis C; Lung Transplant
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lung Transplant (Experimental): Patients will be transplanted with HCV positive lung. Recipients whom test positive for HCV viremia for 2 consecutive tests at any point will complete 12 weeks of Epclusa (Sofosbuvir/velpatasvir).
  Interventions: Drug: Epclusa

INTERVENTIONS:
Drug: Epclusa — Patients testing positive for HCV viremia will receive 12 weeks of Epclusa.
  Other Names: Procedure; Sofosbuvir/velpatasvir

SUMMARY:
To perform a study (20 patients) utilizing Hepatitis C positive (HCV Ab+/NAT -) donor lungs for hepatitis C negative recipients with post-operative surveillance and treatment only if a recipient infection occurs.

DETAILED DESCRIPTION:
The investigators are proposing a study of efficacy, in which positive donors will be used for HCV negative patients. Following lung transplantation patients will undergo HCV antibody, virus PCR, and liver function testing. Recipients whom test positive for HCV viremia for 2 consecutive tests at any point will complete 12 weeks of Sofosbuvir/velpatasvir therapy.

This initial study would enroll 20 patients and utilize donors that are young, otherwise healthy whom are Hepatitis C antibody positive but Nucleic Acid Amplification Testing (NAT) negative (HCV Ab+/NAT-). The recipients would be limited to those patients who have previously consented to receive a high risk lung transplant, consented to participant in this study, and who are physiologically optimized for transplantation (e.g., low risk for lung transplantation).

ELIGIBILITY:
Inclusion Criteria:

* Patients who sign the informed consent for this study
* Patients whom agree to receive a PHS high risk organ
* Patients listed for heart transplantation
* Age 18-65

Exclusion Criteria:

* Patients who do not sign informed consent for this study
* HIV Seropositivity
* HBV Seropositivity (HBcAb and/or HBsAg positive)
* Abnormal liver enzymes - 3 times the normal liver function values (Bilirubin, INR, AST, ALT)
* Acute or chronic renal insufficiency (creatinine clearance <50 ml/min) or history of dialysis
* Patients on ECMO
* Respiratory insufficiency requiring mechanical respiratory support (ventilator, BiPAP)
* Liver insufficiency
* Prior history of hepatitis C
* Allergy to Sofosbuvir/velpatasvir
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
HCV Viremia | at 2 years
  Incidence of HCV Viremia
Seroconversion | at 2 years
  Rate of HCV seroconversion
Liver Function Testing | at 2 years
  Assessment of Hepatic function
Survival | at 2 years
  Survival rates

SECONDARY OUTCOMES:
Rejection | at 2 years
  The incidence of rejection
Waitlist | at 2 years
  Time on waitlist will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Sanchez, MD, Principal Investigator — Assistant Professor of Surgery/University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sofosbuvir — https://druginfo.nlm.nih.gov/drugportal/name/Sofosbuvir
- See also: Drug Information — https://clinicaltrials.gov/ct2/info/fdalinks